CLINICAL TRIAL: NCT03853720
Title: A Pilot Study Evaluating Efficacy and Safety of Combined and Simultaneous Balloon-occluded Retrograde Transvenous and Endoscopic Obliteration of High-risk Gastric Varices
Brief Title: Combined and Simultaneous Approach for the Treatment of High-risk Gastric Varices Using B-RTO and EVO
Acronym: BeRTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Alban Denys, Full Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-02183
Record Dates: First submitted 2019-02-20; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Gastric Varices Bleeding; Gastric Varix
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): combined and simultaneous balloon-occluded retrograde transvenous and endoscopic obliteration of high-risk gastric varices
  Interventions: Procedure: balloon-occluded retrograde transvenous and endoscopic obliteration of high-risk gastric varices

INTERVENTIONS:
Procedure: balloon-occluded retrograde transvenous and endoscopic obliteration of high-risk gastric varices — Catheterization of the left renal vein and the inferior diaphragmatic vein and occlusion with a balloon placed in the distal portion of this vein.
  Endoscopic access to the gastric cavity, gastric varices identification and flow measurement, including velocity, by endoscopic Doppler ultrasound (US). The balloon in the draining vein will be inflated and the velocity will be reassessed. Endoscopic puncture of the varices will be done and the embolization will be conducted under balloon-occlusive conditions (Injection of Cyanoacrylate: Lipiodol mixture 1:1 slowly and gradually). Balloon will be kept inflated and a microcatheter will be used through its lumen inside the variceal bed to inject occlusive agent (cyanoacrylate) mixed with Lipiodol.
  At the end of the procedure an occlusion device (plug amplatzer 2) will be placed.

SUMMARY:
The aim of this pilot study is to evaluate the efficacy and safety of combined and simultaneous endoscopic variceal obliteration together with balloon occluded-retrograde transvenous obliteration (B-RTO) for the treatment of high-risk gastric varices

DETAILED DESCRIPTION:
Although less frequent than esophageal varices, gastric varices constitute a severe and potentially life threatening complication of portal hypertension. Various methods have been described to treat gastric varices, including endoscopic and interventional radiology techniques. Endoscopic variceal obliteration (EVO) is currently considered as standard of care for the treatment of gastric varices in most centers. However, this technique is associated with significant rebleeding rates and incomplete obliteration is observed in about 50% of patients. Alternatively, few centers also use an interventional radiology technique, called balloon-occluded retrograde transvenous obliteration (B-RTO) to treat gastric varices, which has been shown to be associated with less recurrence of gastric varices and high rates of eradication of about 90%. Both techniques have their inherent weaknesses, such as frequent incomplete eradication of varices and thromboembolic events for EVO, while data suggest that B-RTO may aggravate esophageal varices.

The aim of this pilot study is to evaluate the efficacy and safety of combined and simultaneous endoscopic variceal obliteration together with (modified) B-RTO. Stopping the outflow of gastric varices by endovascular balloon occlusion may allow better endoscopic visualization, blood stagnation and thus eradication of varices, while preventing thromboembolic events. Furthermore, during study follow-up, the eradication rates and recurrence of varices, short-term and long term complications, effects of the procedure on portal pressures/hemodynamics and liver function will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent as documented by signature (Appendix "Fiche d'information aux patients et formulaire de consentement éclairé")
2. Patients with endoscopically proven high-risk (diameter >2 cm, mosaic gastropathy, red spots or signs of previous bleeding) and GOV2, IGV1 and IGV2 type of gastric varices (according to Sarin classification)
3. Portal hypertension secondary to cirrhosis
4. Age >18

Exclusion Criteria:

1. Acute gastric or esophageal varice bleeding
2. GOV1 varices according to Sarin classification
3. Hemodynamic instability
4. Uncompensated cirrhosis
5. Contraindication to general anesthesia
6. Contraindication to CT-scan/angiography (impaired kidney function, allergy to iodine based contrast)
7. Allergy to cyanoacrylate, drugs or material used during procedures
8. Absence of gastro-renal shunt
9. Pregnancy
10. Participation to another study involving ionizing radiation (dose superior to 5mSV) without direct benefice for patient during the 12 last months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Gastric varice eradication following intervention (at 4 weeks) | 4 weeks
  Gastric varice eradication following intervention (at 4 weeks) assessed by esophagogastroduodenoscopy (complete eradication or incomplete eradication)

SECONDARY OUTCOMES:
Gastric varice eradication following intervention | 12 weeks
  Gastric varice eradication following intervention (at 12 weeks) assessed by esophagogastroduodenoscopy (complete eradication or incomplete eradication)
Recurrence of gastric varices | 4 weeks
  Recurrence of gastric varices (defined as recurrence of gastric varices after complete eradication (at 4 weeks))
Bleeding rates following procedure | 2 years
  Bleeding rates following procedure (% of patients that had a bleeding at 2 years of follow-up following eradication and mean time to bleeding after procedure)
Effect of procedure on esophageal varices | 2 years
  Effect of procedure on esophageal varices. Classification of "Paquet" with evaluation before procedure and at 2 years after procedure (Paquet Grade 1 to 4)
Effect of procedure on portal pressures | 3 months
  Effect of procedure on portal pressures at 3 months assessed by endovascular hepatic pressure measurment (and compared with pressure before procedure).
Effect of procedure on liver function | 2 years
  Effect of procedure on liver function and cirrhosis assessed by CHILD-PUGH score ((albumin (g/l) : >35 = 1 point ; 28-35 = 2 points ; <28 = 3 points); (total bilirubin (umol/l)<34 = 1 point ; 34-50 = 2 points; >50 = 3 points); (INR : <1.7 = 1 point; 1.71-2.30 = 2 points; >2.30 = 3 points), (Ascites: none = 1 point; mild = 2 points, moderate/severe= 3 points); (Hepatic Encephalopathy: none = 1 point; Grade I-II = 2 points; Grade III-IV = 3 points). Total score : 5-6 = A ; 7-9 = B; 10-15 = C.
Description of procedural complications | 2 years
  Description of procedural complications (bleeding, pulmonary embolism)
Description of pre-treatment variceal anatomy/classification | 1 day
  Description of pre-treatment variceal anatomy/classification according to Sarin Classification

CONTACTS AND LOCATIONS:
Overall Officials: Alban Denys, MD, Principal Investigator — Full Professor

IPD SHARING:
Plan to Share IPD: No